CLINICAL TRIAL: NCT07177053
Title: Comparative Clinical Evaluation of Remineralization of Molar Incisor Hypomineralization Using Hydroxyapatite vs. Fluoride Toothpaste
Brief Title: Hydroxyapatite vs Fluoride Toothpaste for MIH Remineralization
Acronym: MIH-CARE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dubai Health (Other Government)
Responsible Party: Principal Investigator, Shaima Buhamer, Specialist Pediatric Dentist, Dubai Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Not yet issued
Record Dates: First submitted 2025-08-30; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Molar Incisor Hypomineralisation
Keywords: Molar Incisor Hypomineralization (MIH); Child; Remineralization; Hydroxyapatite Toothpaste; Fluoride Toothpaste; Quantitative Light-Induced Fluorescence(QLF)
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydroxyapatite tooth paste [ HAP] (study group) (Active Comparator)
  Interventions: Drug: non fluoridated hydroxyapatite tooth paste (KAREX KINDER tooth paste)
- Fluoride-containing tooth paste [1450ppm fluoride] (control group) (Active Comparator)
  Interventions: Drug: fluoridated toothpaste (Colgate Total PROTECTION ACTIVE)

INTERVENTIONS:
Drug: non fluoridated hydroxyapatite tooth paste (KAREX KINDER tooth paste) — arm 1 : hydroxyapatite tooth paste [ HAP] (study group): assessment will involve Quantitative Light-Induced Fluorescence- QLF at baseline, 3, 6, 9, and 12 months. The images were analyzed using a commercial software program (Inspektor QLF 1.97, Inspektor Research Systems, Amsterdam, The Netherlands) to determine the change in fluorescence
  (ΔF, %) and extension of the lesion (area; mm2).
  Arms: hydroxyapatite tooth paste [ HAP] (study group)
Drug: fluoridated toothpaste (Colgate Total PROTECTION ACTIVE) — Arm 2 :Fluoride-containing tooth paste [1450ppm fluoride] (control group):
  assessment will involve Quantitative Light-Induced Fluorescence- QLF at baseline, 3, 6, 9, and 12 months. The images were analyzed using a commercial software program (Inspektor QLF 1.97, Inspektor Research Systems, Amsterdam, The Netherlands) to determine the change in fluorescence (ΔF, %) and extension of the lesion (area; mm2).
  Arms: Fluoride-containing tooth paste [1450ppm fluoride] (control group)

SUMMARY:
Molar Incisor Hypomineralization (MIH) is a common developmental enamel defect affecting children, particularly in Dubai, where it contributes to hypersensitivity, esthetic concerns, plaque accumulation, and increased caries risk. These complications often lead to premature tooth extraction and orthodontic issues, negatively impacting children's oral health-related quality of life.

This randomized, open-label clinical trial aims to compare the remineralization efficacy of a fluoride-free hydroxyapatite toothpaste with a conventional fluoride toothpaste in children aged 6-12 years diagnosed with mild to moderate MIH.

Participants will be recruited from Dubai Health pediatric dental clinics, with inclusion criteria requiring at least one affected permanent molar or incisor, good general health, parental informed consent, and the child's assent. Children with systemic conditions affecting enamel or recent use of desensitizing treatments will be excluded.

Primary outcome assessment will involve Quantitative Light-Induced Fluorescence-QLF at baseline, 3, 6, 9, and 12 months. The images were analyzed using a commercial software program (Inspektor QLF 1.97, Inspektor Research Systems, Amsterdam, The Netherlands) to determine the change in fluorescence (ΔF, %) and extension of the lesion (area; mm2).

Secondary outcome measures will include enamel fluorescence readings using the DIAGNOdent Pen. After prophylaxis and air-drying, three readings per lesion will be recorded, with mean and peak values analyzed to monitor mineralization. Hypersensitivity in MIH-affected teeth will be assessed using air stimulus (Schiff scale) and Visual Analogue Scale (VAS) at baseline, 3, 6, 9, and 12 months. Oral health-related quality of life (OHRQoL) will be measured using age-appropriate validated questionnaires to evaluate the impact of MIH and treatment over time.

This study also responds to growing parental concerns about fluoride exposure and the demand for safer, fluoride-free alternatives. By evaluating the clinical effectiveness of hydroxyapatite toothpaste, the trial aims to inform evidence-based preventive strategies for MIH management. The findings may guide clinical practice and public health recommendations, ultimately improving oral health outcomes for affected children.

DETAILED DESCRIPTION:
Molar Incisor Hypomineralization (MIH) affects approximately 13-14% of children globally. It is a developmental enamel defect with multifactorial etiology, including perinatal and early childhood illnesses. Clinically, MIH leads to hypersensitivity, enamel breakdown, and increased caries risk, significantly impacting oral health-related quality of life. Remineralization strategies using fluoride and biomimetic agents like hydroxyapatite (HAP) have shown promise. HAP offers comparable efficacy to fluoride with added benefits and fewer risks.

Molar incisor hypomineralization (MIH) is a qualitative enamel defect affecting up to 14% of children globally. It is associated with enamel breakdown, hypersensitivity, and increased caries risk. Fluoride is widely used for remineralization but carries risks like fluorosis. Hydroxyapatite (HAP), a biomimetic agent, has shown comparable efficacy in caries prevention and remineralization. However, there is a lack of in vivo clinical trials comparing HAP and fluoride for MIH management in children. This study addresses the need for safer, effective alternatives to fluoride in pediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

* at least one affected permanent molar or incisor
* good general health
* parental informed consent, and the child's assent

Exclusion Criteria:

* Patients with systemic conditions affecting enamel or recent use of desensitizing treatments.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Enamel remineralization - Fluorescence Change (ΔF, %) | 3,6,9,12 months
  Unit of measure: Percent change in fluorescence intensity (ΔF, %)
  Measurement tool/method: Quantitative Light-Induced Fluorescence (QLF) imaging; images analysed with Inspektor QLF software (v1.97).
Enamel remineralization - Lesion Area (mm²) | Baseline, 3, 6, 9, and 12 months.
  Unit of measure: Lesion surface area (mm²)
  Measurement tool/method: Quantitative Light-Induced Fluorescence (QLF) imaging; images analysed with Inspektor QLF software (v1.97).

SECONDARY OUTCOMES:
Enamel fluorescence (adjunct) | 3,6,9,12 months
  Unit of measure: DIAGNOdent value (device units; 0-99) - numeric reading reported by the DIAGNOdent Pen (mean and peak values per lesion).
  Measurement tool / method: DIAGNOdent Pen fluorescence readings (three readings per lesion after prophylaxis and air-drying; report mean and peak).
Hypersensitivity- Schiff Cold Air Sensitivity Scale Score | Baseline, 3, 6, 9, and 12 months.
  Unit of measure: Ordinal score (0-3) per tooth
  Scale description: Schiff Cold Air Sensitivity Scale; minimum = 0 (no response), maximum = 3 (severe painful response).
  Interpretation: Higher scores indicate worse hypersensitivity.
  Measurement tool/method: 1-second air blast (40-65 psi, 1 cm distance) applied to the affected tooth; response scored by examiner.
Visual Analogue Scale (VAS) for Hypersensitivity | Baseline, 3, 6, 9, and 12 months.
  Unit of measure: Continuous score (0-10 cm)
  Scale description: Visual Analogue Scale; minimum = 0 cm (no pain), maximum = 10 cm (worst imaginable pain).
  Interpretation: Higher scores indicate worse hypersensitivity.
  Measurement tool/method: Immediately after the air stimulus, the child self-reports hypersensitivity by marking on a 10 cm VAS line.
Oral health-related quality of life (OHRQoL) | Baseline and 6 months
  Unit of measure: Total CPQ score (numeric sum); change in total and domain scores from baseline.
  Measurement tool/method: Child Perceptions Questionnaire (CPQ), age-appropriate validated versions (e.g., CPQ8-10, CPQ11-14), using validated Arabic translations where applicable.
  Scale description:
  CPQ8-10: 25 items, total score range = 0 to 100.
  CPQ11-14: 37 items, total score range = 0 to 148.
  Higher scores indicate worse oral health-related quality of life (more negative impact).